CLINICAL TRIAL: NCT03857841
Title: A Safety Study of Intravenous Infusion of Bone Marrow Mesenchymal Stem Cell-derived Extracellular Vesicles (UNEX-42) in Preterm Neonates at High Risk for Bronchopulmonary Dysplasia
Brief Title: A Safety Study of IV Stem Cell-derived Extracellular Vesicles (UNEX-42) in Preterm Neonates at High Risk for BPD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was discontinued due to a business decision; no safety concerns were noted.
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UNX-BP-101
Record Dates: First submitted 2019-02-20; First posted 2019-02-28 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary Dysplasia; Mesenchymal Stem Cell-derived Extracellular Vesicles; Preterm Neonates
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 20 pmol phospholipid/kg body weight (Experimental): UNEX-42 administered at 20 pmol phospholipid/kg body weight
  Interventions: Biological: UNEX-42
- 60 pmol phospholipid/kg body weight (Experimental): UNEX-42 administered at 60 pmol phospholipid/kg body weight
  Interventions: Biological: UNEX-42
- 200 pmol phospholipid/kg body weight (Experimental): UNEX-42 administered at 200 pmol phospholipid/kg body weight
  Interventions: Biological: UNEX-42
- Placebo (Placebo Comparator): Phosphate-buffered saline
  Interventions: Biological: Phosphate-buffered saline

INTERVENTIONS:
Biological: UNEX-42 — UNEX-42 is a preparation of extracellular vesicles that are secreted from human bone marrow-derived mesenchymal stem cells suspended in phosphate-buffered saline.
  Arms: 20 pmol phospholipid/kg body weight; 200 pmol phospholipid/kg body weight; 60 pmol phospholipid/kg body weight
Biological: Phosphate-buffered saline — Phosphate-buffered saline
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
A multicenter, placebo-controlled, randomized, dose escalation, safety, and tolerability study of UNEX-42 in infants born at <27 weeks of gestational age (GA) at high risk for bronchopulmonary dysplasia (BPD).

DETAILED DESCRIPTION:
The study was discontinued by the Sponsor on 24 February 2021 due to a business decision, not related to reasons of safety or efficacy. Only data listings were created; no summary or inferential analyses were performed.

Subjects were assessed during Screening and Baseline (prior to randomization) for eligibility in the study. Subjects then received a single IV dose of UNEX-42 at 20 pmol phospholipid/kg body weight, or placebo. After randomization, subjects were monitored in the hospital through 40 Weeks postmentrual age (PMA) or the time of hospital discharge (whichever came first).

The following efficacy and safety assessments occurred during the course of the study:

Efficacy Assessments: incidence and severity of BPD, duration of hospitalization, duration of mechanical ventilation, duration of supplemental oxygen therapy, duration of postnatal steroids, tracheal aspirate inflammatory biomarkers, and Respiratory Severity Score.

Safety Assessments: physical examination, vital signs, adverse events, predefined complications of prematurity, clinical laboratory parameters, and chest x-ray.

Dose administration for Cohort 1 occurred so that there was an observational period of 3 days between dosing the first, second, and third subject to assure the opportunity for safety assessments in at least 1 subject on active treatment. In addition, enrollment between cohorts was to be paused for data review by a Data Monitoring Committee to evaluate the data available after each of the first 2 cohorts were enrolled.

Subjects that completed the Post-treatment Phase (including those that were discharged from the hospital prior to 40 Weeks PMA) continued into the Long-term Outcome Phase and were assessed through 1 year of corrected age.

ELIGIBILITY:
Inclusion Criteria:

1. Infant whose postnatal age was 3 to 14 days
2. Subjects met the following oxygen and birth weight criteria based on gestational age: 23 weeks to 24 weeks 6 days (any birth weight, any oxygen requirement) or 25 weeks to 26 weeks 6 days (fraction of inspired oxygen [FiO2] ≥35% [sustained for >2 hours] at any point during postnatal Days 1 to 14 AND birth weight ≤750 g)
3. Endotracheally intubated and receiving mechanical ventilation at the time of Screening and randomization.
4. Not expected to be extubated within the next 24 hours after randomization.
5. The subject had a parent/guardian who gave written informed consent.

Exclusion Criteria:

1. Had a congenital heart defect, except for PDA, atrial septal defect or a small/moderate, restrictive ventricular septal defect.
2. Had a serious malformation of the lung, such as pulmonary hypoplasia/aplasia, congenital diaphragmatic hernia, or any other congenital lung anomaly.
3. Was being treated with inhaled nitric oxide.
4. Had a known chromosomal abnormality (eg, Trisomy 18, Trisomy 13, or Trisomy 21) or a severe congenital malformation (eg, hydrocephalus and encephalocele, trachea-esophageal fistula, abdominal wall defects, and major renal anomalies).
5. Had a known severe congenital infectious disease (ie, herpes, toxoplasmosis rubella, syphilis, human immunodeficiency virus, cytomegalovirus, etc).
6. High clinical suspicion of active systemic infection, severe sepsis, or septic shock during Screening.
7. Underwent a surgical procedure (requiring admission to an operating room) within 72 hours before randomization or who was anticipated to have a surgical procedure (requiring admission to an operating room) within 72 hours before or following randomization.
8. Had a Grade 3 or 4 intracranial hemorrhage.
9. Had active pulmonary hemorrhage.
10. The subject was currently participating in any other interventional clinical study.
11. The subject was, in the opinion of the Investigator, so ill that death was inevitable, or was considered inappropriate for the study for any reason(s) other than those listed above.

Ages: 3 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-05-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Colorado Hospital, Aurora, Colorado
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 20 Pmol Phospholipid/kg Body Weight | 60 Pmol Phospholipid/kg Body Weight | 200 Pmol Phospholipid/kg Body Weight | Placebo
Started | 2 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 1
Not Completed | 2 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Study Terminated by Sponsor | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects randomized and received clinical study material
Groups:
- Total: Total of all reporting groups
Arm/Group | 20 Pmol Phospholipid/kg Body Weight | 60 Pmol Phospholipid/kg Body Weight | 200 Pmol Phospholipid/kg Body Weight | Placebo | Total
Number analyzed (Participants) | 2 | 0 | 0 | 1 | 3
Age, Customized [Number; unit: participants]
  Postnatal Age - 5 Days | 0 |  |  | 1 | 1
  Postnatal Age - 7 Days | 1 |  |  | 0 | 1
  Postnatal Age - 12 Days | 1 |  |  | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 1 | 3
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 |  |  | 0 | 1
  Not Hispanic or Latino | 1 |  |  | 1 | 2
  Unknown or Not Reported | 0 |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  |  | 0 | 0
  Asian | 0 |  |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0 | 0
  Black or African American | 2 |  |  | 1 | 3
  White | 0 |  |  | 0 | 0
  More than one race | 0 |  |  | 0 | 0
  Unknown or Not Reported | 0 |  |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  |  | 1 | 3
Gestation Age at Birth [Number; unit: participants]
  23 Weeks/0 Days | 0 |  |  | 1 | 1
  24 Weeks/1 Day | 1 |  |  | 0 | 1
  24 Weeks/5 Days | 1 |  |  | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events During the Post-treatment Phase (Safety and Tolerability)
Description: The safety and tolerability of UNEX-42 in subjects with BPD was evaluated by the number of subjects with treatment-emergent adverse events, including death, computed by dose cohort and overall during the Post-treatment Phase.
Time Frame: From Day 1 to 40 Weeks Post-menstrual Age or Hospital Discharge, whichever came first
Population: All subjects randomized and received clinical study material.
Measure: Count of Participants; unit: Participants
Arm/Group | 20 Pmol Phospholipid/kg Body Weight | 60 Pmol Phospholipid/kg Body Weight | 200 Pmol Phospholipid/kg Body Weight | Placebo
Number analyzed (Participants) | 2 | 0 | 0 | 1
Participants | 2 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From Day -2 to 40 Weeks Post-menstrual Age or Hospital Discharge, whichever came first
Description: Specific complications of prematurity were assessed from Screening to 40 Weeks PMA/Hospital Discharge. Complications of prematurity were only recorded as an AE or SAE if the event was unusual with respect to intensity, frequency, duration as compared with symptoms in the subject's medical history, or if there was a reasonable possibility that the event was caused by the study drug. Congenital disorders were recorded as medical history, even if diagnosed after the subject had entered the study.
Arm/Group | 20 Pmol Phospholipid/kg Body Weight | 60 Pmol Phospholipid/kg Body Weight | 200 Pmol Phospholipid/kg Body Weight | Placebo
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/0 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/0 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0 | 0/0 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 Pmol Phospholipid/kg Body Weight (N=2) | 60 Pmol Phospholipid/kg Body Weight (N=0) | 200 Pmol Phospholipid/kg Body Weight (N=0) | Placebo (N=1)
Necrotizing colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 Pmol Phospholipid/kg Body Weight (N=2) | 60 Pmol Phospholipid/kg Body Weight (N=0) | 200 Pmol Phospholipid/kg Body Weight (N=0) | Placebo (N=1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Generalized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Beta hemolytic streptococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any interim results of the study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.

DOCUMENTS (2):
  • Study Protocol (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT03857841/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-11): https://cdn.clinicaltrials.gov/large-docs/41/NCT03857841/SAP_001.pdf